CLINICAL TRIAL: NCT01131689
Title: Phase 1 Trial of S-1 in Combination With Sorafenib for Patients With Advanced Hepatocellular Carcinoma
Brief Title: Trial of S-1 in Combination With Sorafenib for Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-10-009
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: metastatic HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sorafenib, TS-1 — D1-14 S-1 dose of level 1/2/3/4 D1-21 Sorafenib 400mg twice daily Every 3 weeks-cycle

SUMMARY:
In preclinical studies, 5-fluorouracil, one of the active metabolites of S-1, showed synergistic effect to sorafenib in human colon carcinoma cell lines. Therefore, sorafenib combined with S-1 might be more effective treatment for patients with advanced HCC than sorafenib monotherapy. The investigators propose to conduct a phase I study to determine maximal tolerated dose (MTD) of S-1 in combination with fixed dose of sorafenib in patients with advanced HCC

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed hepatocellular carcinoma (HCC) or a combination of radiologically compatible finding to HCC, alpha-fetoprotein>400ng/mL and liver cirrhosis
2. Inoperable disease as defined by

   1. Localized disease in a portion of the liver that doses not allow the possibility of complete surgical removal of the tumor with a clear resection margin OR
   2. Presence of extra-hepatic disease OR
   3. Main portal vein or hepatic vein involvement (invasion or tumor thrombus) OR
   4. The HCC must not be amenable to intra-arterial therapy or local ablative therapy
3. Minimum life expectancy of 12 weeks
4. Age>18 years.
5. ECOG Performance Status of 0-1
6. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   1. Hemoglobin>9.0 g/dl
   2. Absolute neutrophil count (ANC) >1,500/mm3
   3. Platelet count > 75,000/μl
   4. Total bilirubin < 1.5 times the upper limit of normal
   5. ALT and AST <5 x upper limit of normal
   6. Albumin >= 3g/dL
   7. PT-INR/PTT <1.5 x upper limit of normal
   8. Serum creatinine < 1.5 x upper limit of normal or Creatinine clearance >=50mL/min
7. Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

1. Decompensated cirrhosis or stage C according to the Child-Pugh Classification
2. Chemo-embolization within 8 weeks of inclusion
3. Other concomitant anticancer agent, including Tamoxifen and Interferon
4. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
5. History of HIV infection
6. Active clinically serious infections (> grade 2 CTCAE version 3.0)
7. Symptomatic metastatic brain or meningeal tumors
8. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
9. History of organ allograft
10. Patients with evidence or history of bleeding diathesis
11. Patients undergoing renal dialysis
12. Radiotherapy during study or within 4 weeks of start of study drug.
13. Major surgery within 4 weeks of start of study
14. Autologous bone marrow transplant or stem cell rescue within 4 months of study
15. Prior exposure to the study drug.
16. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial (and men for at least 3 months after last administration of study medication).
17. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
18. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
19. Patients unable to swallow oral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
MTD | 1 year
  Primary objectives:
  1. To determine maximal tolerated dose (MTD) of S-1 combined with fixed dose of sorafenib 400mg twice daily.
  Secondary objectives:
  1. To evaluate toxicity profiles and dose-limiting toxicity (DLT)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea